CLINICAL TRIAL: NCT00892827
Title: The Efficacy and Safety of Combined Treatment With Fresh Frozen Plasma and Rituximab (Mabthera) in Patients With Advanced Refractory Chronic Lymphocytic Leukemia. Single-arm Phase II Study. Analysis of Complement Activation Pathways.
Brief Title: Combined Treatment With Fresh Frozen Plasma and Rituximab (Mabthera) in Patients With Advanced Refractory Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr. Klepfish A., Director of Blood Bank, Wolfson Medical Center, Holon, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK- 01
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Refractory Chronic Lymphocytic Leukemia
Keywords: Rituximab; Mabthera; FFP; Fresh Frozen Plasma; CLL; Complement; Response; Overall response rate of FFP+Rituximab combined therapy; Analysis of complement activation pathways prior to, during and; after the study treatment.; Time to disease progression; Time to re-treatment (See Appendix I).; Safety of the combination treatment of FFP and RTX.
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental): Rituximab
  Interventions: Drug: Rituximab (Mabthera) , FFP (Fresh Frozen Plasma)

INTERVENTIONS:
Drug: Rituximab (Mabthera) , FFP (Fresh Frozen Plasma) — Rituximab (375 mg/m2) with FFP will be given every two weeks

SUMMARY:
Chronic lymphocytic leukemia (CLL), an indolent disease of mature-looking B lymphocytes, is the most common leukemia in Israel and the Western world. The disease is associated with considerable morbidity and mortality, and is currently incurable. Rituximab (Mabthera) is a chimeric monoclonal antibody directed against CD20 antigen, present exclusively on B lymphocytes. Treatment with Rituximab is widely used in indolent B cell malignancies. However, the administration of Rituximab in CLL patients yields less successful results than in other indolent B cell malignancies, and even responding patients may become refractory. We hypothesized that the abnormalities in the complement system identified in CLL underlie the suboptimal response to Rituximab, since complement-dependent cell cytotoxicity is a major mechanism of Rituximab action. Following patient consent and Institutional Review Board approval, standard-dose Rituximab (375 mg/m2) will be administered, preceded by 2 units of FFP. This treatment will be repeated every 1-2 weeks for 4-6 cycles. The clinical and laboratory parameters, as well as adverse drug events, will be monitored.

DETAILED DESCRIPTION:
Indolent B cell Non-Hodgkin's lymphoma patients show good responses to Rituximab, administered either alone or preferably with standard chemotherapy. The response to Rituximab of patients with CLL is inferior in comparison to other indolent B cell malignancies. The therapeutic approach of combining treatments with Rituximab and fresh frozen plasma (FFP) used by us first in one case and following the impressive response - in additional 2 patients, was undertaken on the basis of two observations.

We assumed, that the addition of FFP to Rituximab treatment would increase and/or restore the efficacy of Rituximab in advanced CLL patients that are resistant to therapy by correcting their abnormal complement system thus allowing improved complement activation and increase anti-leukemic activity.

The major aims of the study are: (1) To establish the efficacy of the combination of FFP and RTX as determined by response rate. (2) To elucidate the effector mechanism responsible for the efficacy of the FFP-Rituximab combination. The secondary aims of the study are (1) To establish the response duration of the combination of FFP and RTX as determined by time to progression. and time to re treatment (2) To determine the safety of the combined treatment.

The study is designed as a single-arm, phase II study evaluating the efficacy and safety of combined treatment with FFP and RTX in advanced refractory chronic lymphocytic leukemia, along with an analysis of the complement system associated parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: advanced (Rai stage ≥2 or symptomatic stage 1) CLL Resistant to or relapsing after treatment with Fludarabine and/or Rituximab
* Lymphocyte count of 100,000 cells/mcl or higher.
* Time from last anti-leukemia treatment: 1 month or more
* Age: male or female over 18 years of age.
* Informed consent - obtained

Exclusion Criteria:

* Lack of one or more of the inclusion criteria
* Known sensitivity to human plasma
* Known sensitivity to Rituximab (Mabthera)
* Active second malignant disease (other than non-melanoma skin cancer) < 2 years prior to the study
* Active infectious disease < 1 month prior to the study
* Hepatitis B serology: Hepatitis B surface antigen - positive
* Renal function: Creatinin > 3 mg/dL
* Liver function: Liver enzymes less than x2 of the normal values
* Performance status: ECOG performance status 4
* Use of other investigational agent < 30 days ago
* Known poor adherence to treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To establish the efficacy of the combination of FFP and RTX as determined by response rate. Complete/Partial Response includes parameters: Physical Exam,Symptoms,Lymphocytes, Neutrophils, Platelets,Hb (g/dL),Bone marrow lymph | 3 months

SECONDARY OUTCOMES:
Time to disease progression | 6-12 months
Time to re-treatment | 6-12 months
Safety of the combination treatment of FFP and RTX | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson MC, Holon, Holon, Israel